

## **Study Protocol**:

This will be a prospective study to be performed at Le Bonheur Children's Hospital. Total study duration for each patient will be 1 year. All patients enrolled in the study will be on the same folic acid dose of 800mcg. Folate levels will be obtained from each patient at the onset of the study, and these will act as the controls. Each patient will then be placed on weekly folic acid dosing, and repeat folate levels will be obtained at 6-month intervals until conclusion of the study.